CLINICAL TRIAL: NCT00526656
Title: Phase II Single Arm, Open Label, Single Institution Study of Neoadjuvant Sunitinib (SUTENT) in Patients With Muscle-Invasive Locally Advanced Transitional Cell Carcinoma of the Bladder
Brief Title: Sunitinib in Treating Patients With Locally Advanced Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE24806; P30CA043703 (NIH); GA6180CV (Other Grant/Funding Number: Pfizer-GA6180CV)
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sunitinib; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sunitinib malate (Experimental): Drug
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — 50mg PO daily 4 weeks on -2 weeks off
  Other Names: Drug

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sunitinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying the side effects and how well sunitinib works in treating patients with locally advanced bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the pathologic complete response rate of sunitinib malate in patients with muscle-invasive locally advanced transitional cell carcinoma (TCC) of the bladder.
* To evaluate the safety and tolerability of sunitinib malate administered prior to radical cystectomy, including surgical outcome and surgical complications.

Secondary

* To determine the clinical effects of sunitinib malate administered prior to radical cystectomy and bilateral lymph node dissection, including overall response rate using RECIST defined criteria, cytology, and histologic appearance of surgical specimen as well as time to progression.

Tertiary

* To assess pre-treatment tissue baseline angiogenic markers and to evaluate the magnitude of the difference among these variables with post-treatment tumor tissue after neoadjuvant sunitinib malate.
* To evaluate the effects of sunitinib malate on immunosuppressive regulatory T cells.

OUTLINE: Patients receive oral sunitinib malate once daily in weeks 1-4 (1 course). Patients undergo restaging within 1 week prior to surgery and then undergo radical cystectomy and bilateral lymph node dissection on day 42. Patients achieving a complete pathologic response at the time of surgery may receive 6 more courses of adjuvant sunitinib malate beginning 28 days after surgery at the discretion of the treating physician. Patients found to have high-risk features (i.e. pT3 or greater tumor and evidence of disease in any of the lymph nodes resected) are offered standard adjuvant systemic chemotherapy at the discretion of the treating physician.

Tumor tissue from pretreatment biopsy and radical cystectomy will be tested for VEGFR-1, VEGFR-2 and PDGF-R expression by IHC. Samples are also analyzed for quantification of cell proliferation and apoptosis and immunosuppressive regulatory T cells (T-reg) and T-reg functions.

After completion of study treatment, patients are followed at 28 days after surgery.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histological confirmed transitional cell carcinoma (TCC) of the bladder

  * Patients with mixed tumors (i.e., tumors containing elements of squamous cell or adenocarcinoma) are eligible
  * Patients with pure non-transitional cell carcinomas are not eligible
* Meets 1 of the following staging criteria:

  * Tumors ≥ cT2

    * Patients with cT2 lesions must have either a bulky or fixed lesion at the time of physical examination and/or scans
  * Any cT stage with nodal-positive disease (documented by scans)

    * Patients with (+) N1-N3 disease are eligible
* Candidate for radical cystectomy in ≥ 8 weeks while neoadjuvant sunitinib malate is administered

Exclusion criteria:

* Any evidence of distant metastasis (excluding pelvic or retroperitoneal lymph nodes)

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status (PS) 0-1 (Karnofsky PS greater than 70%)
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Hemoglobin ≥ 8.5 g/dL
* Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN)
* AST and ALT ≤ 3.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 10 times ULN in presence of bone metastasis)
* Serum calcium ≤ 12 mg/dL
* Creatinine ≤ 1.5 times ULN
* INR ≤ 1.5 (except for patients receiving warfarin therapy)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Disease-free of prior malignancies for ≥ 5 years except for currently treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix

Exclusion criteria:

* NCI CTCAE grade 3 hemorrhage within 4 weeks of starting study treatment
* Any of the following within 6 months prior to study drug administration:

  * Myocardial infarction
  * Severe/unstable angina
  * Coronary/peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
* Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥ 2, atrial fibrillation of any grade, or prolongation of the QTc interval to > 450 msec for males or > 470 msec for females
* Hypertension that cannot be controlled by medications
* Known HIV or AIDS-related illness
* Infectious hepatitis type A, B, or C
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Other systemic chemotherapy must have been completed at least 5 years prior to enrollment
* No prior systemic chemotherapy for bladder cancer
* No other approved or investigational anticancer treatment will be permitted during the study period, including chemotherapy, biological response modifiers, hormone therapy, surgery, palliative radiotherapy, or immunotherapy
* No other investigational drug may be used during treatment on this protocol
* No concurrent participation in another clinical trial

Exclusion criteria:

* Prior intravesical chemotherapy or immunotherapy
* Prior treatment with any other antiangiogenic therapy (including immunomodulatory agents such as thalidomide and lenalidomide and anti-VEGF therapy with agents such as bevacizumab, sunitinib malate, and sorafenib tosylate)
* Prior surgery, radiotherapy, or systemic therapy within 4 weeks of starting the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A. Garcia, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eleven patients were entered into the trial between 9/07 and 12/09 from medical clinic. Two patients were considered ineligible and received no treatment.
Groups:
- Sunitinib Malate: Drug
  sunitinib malate : 50mg PO daily 4 weeks on -2 weeks off
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 9
Completed | 7
Not Completed | 2
Not completed — Death | 1
Not completed — Refused surgery | 1

BASELINE CHARACTERISTICS:
Population: All participants that were on study.
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 62 [51 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate of Sunitinib
Description: Number of participants who at the time of cystectomy, to have no evidence of tumor grossly and microscopically on routine Hematoxylin and Eosin stain (H&E) (pathologic complete response or P0) will be defined as responders. All cases will be defined as responders (P0) or non-responders based on the presence of residual tumor.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
  Progression (PD): At least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum LD since the treatment started.
Time Frame: at 6 weeks
Population: Participants who completed treatment and surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Evaluate Treatment to Surgical Complication and Morbidity
Description: Determine if surgical morbidity was increased from time of last dose to time of surgery is defined as the number of subjects with increase non-ileus related morbidity due to treatment drug during the 2 week rest period.
Time Frame: following surgery at 6 weeks
Population: Participants who received treatment and surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 7
Participants | 0

3. Secondary Outcome: Time to Progression
Description: Time to progression will be measured as the time from when the patient started treatment to the time the patient is first recorded as having disease progression or the date of death if the patient dies due to causes other than disease progression.
Time Frame: at 4 weeks post-surgery
Population: Data not collected.
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events (SAEs and AEs) collected from consent signed, while on treatment and followed 28 days after the last dose of treatment or until resolved or determined chronic or stable, whichever is later.
Arm/Group | Sunitinib Malate
All-Cause Mortality (participants affected / at risk) | 7/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate (N=9)
Hemoglobin (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Death not associated with CTCAE term - Sudden death (General disorders) | 1
Hemorrhage, GU - Urethra (Renal and urinary disorders) | 1
Hematoma (Vascular disorders) | 1
Infection with no more than Grade 2 ANC: Wound (Infections and infestations) | 1
Edema: limb (General disorders) | 1
Calcium, serum-low (hypocalcemia) (Investigations) | 1
Phosphate, serum-low (hypophosphatemia) (Investigations) | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate (N=9)
Otitis, middle ear (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 6
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 4
Hypertension (Cardiac disorders) | 4
PTT (Partial Thromboplastin Time) (Investigations) | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4
Rigors/chills (General disorders) | 1
Weight loss (General disorders) | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Salivary gland changes/saliva (Gastrointestinal disorders) | 1
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1
Hemorrhage, GU - Bladder (Renal and urinary disorders) | 1
Colitis, infectious (Infections and infestations) | 1
Febrile neutropenia (fever of unknown origin >=38.5; no infection, ANC<1.0x10e9/L) (Infections and infestations) | 1
Edema: limb (General disorders) | 2
Albumin, serum-low (hypoalbuminemia) (Investigations) | 2
Alkaline phosphatase (Investigations) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1
Calcium, serum-high (hypercalcemia) (Investigations) | 1
Calcium, serum-low (hypocalcemia) (Investigations) | 1
Creatinine (Investigations) | 1
Glucose, serum-high (hyperglycemia) (Investigations) | 4
Phosphate, serum-low (hypophosphatemia) (Investigations) | 1
Potassium, serum-high (hyperkalemia) (Investigations) | 1
Sodium, serum-low (hyponatremia) (Investigations) | 2
Mood alteration - Anxiety (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1
Pain - Oral cavity (Gastrointestinal disorders) | 1
Pain - Pain NOS (General disorders) | 1
Pain - Scalp (Skin and subcutaneous tissue disorders) | 1
Pain - Urethra (Renal and urinary disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Urine color change (Renal and urinary disorders) | 1
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 1 — change from baseline
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes